CLINICAL TRIAL: NCT05855343
Title: Exploratory Study of Switching From Combustible Cigarettes to the BIDI E-cigarette
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rose Research Center, LLC (Industry)
Collaborators: Foundation for a Smoke Free World INC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIDI
Record Dates: First submitted 2023-01-25; First posted 2023-05-11 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Smoking Cessation
Keywords: e-cigarette
MeSH Terms: conditions — Smoking Cessation; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BIDI Stick e-cigarette (Experimental)
  Interventions: Other: BIDI Stick e-cigarette

INTERVENTIONS:
Other: BIDI Stick e-cigarette — The BIDI will be dispensed, and subjects will be instructed to use the BIDI as often as they like during the 12 week period, and to switch completely to the BIDI within 1 week. If, however, they do smoke any CC, they will also be instructed to use the BIDI immediately before each CC to relieve their craving as much as possible before smoking their usual brand. The BIDI will also be the first product that they are instructed to use each morning. Smokers will be told to try to completely substitute BIDI for CCs by the end of the first week of use.

SUMMARY:
The aim of this study is to shed light on the importance of nicotine pharmacokinetics in switching to a reduced-harm product by fully matching the nicotine pharmacokinetics of smokers' usual brands of cigarettes.

The primary objective is to ascertain the degree of smoking reduction when smokers attempt to switch to an e-cigarette that matches peak nicotine concentrations of a cigarette.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed the ICF and is able to understand the information provided in the ICF.
2. Is 22 to 65 years of age (inclusive) at screening.
3. Smokes ≥ 10 commercially available CCs per day (no brand restrictions), for the last 12 months.
4. Expired air CO reading of at least 10 ppm as assessed at the screening session.
5. Interested in switching to an electronic cigarette.
6. Willing and able to comply with the requirements of the study.
7. Owns a smart phone with text message and data capabilities compatible with necessary surveys.

Exclusion Criteria:

1. Is unhealthy or cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason) as judged by the Investigator or designated medical staff based on all available assessments from the screening period (e.g., vital signs, physical examination, ECG, concomitant medications and medical history).
2. PHQ-9 score greater than 9, or a score greater than 0 on item #9 ("Thoughts that you would be better off dead, or of hurting yourself in some way") at screening.
3. Planned use of an FDA-approved smoking cessation product during the study.
4. High Blood Pressure (systolic >150 mm Hg, diastolic >95 mm Hg) at screening.
5. Body mass index (BMI) less than 15.0 kg/m2 or greater than 40.0 kg/m2 at screening.
6. Coronary heart disease, structural cardiac disease (including, but not limited to valvular heart disease or cardiac murmurs), cardiac dysrhythmias, syncope, cardiac chest pain, or history of heart attack or heart failure.
7. Has received psychotherapy or behavioral treatments within 30 days of screening, or during the study.
8. Taking antidepressants or psychoactive medications (e.g. antipsychotics, benzodiazepines, hypnotics).
9. Use of any of these products in the past 30 days:

   1. Illegal drugs (or if the urine drug screen is positive for cocaine, THC, amphetamines, phencyclidine (PCP), or opiates without a medical prescription);
   2. Experimental (investigational) drugs that are unknown to participant;
   3. Chronic opiate use.
10. Use of smokeless tobacco (chewing tobacco, snuff), cigars (except for "Black & Mild" cigars or Cigarillos), pipes, hookah, e-cigarettes, nicotine replacement therapy or other smoking cessation treatments within 14 days of screening.
11. Pregnant or nursing (by self-report) or positive pregnancy test.
12. Enrollment is complete.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Degree of Smoking Reduction | After 12 Weeks
  Change in expired air carbon monoxide (CO) at the end of the product use period
Degree of Smoking Reduction | From Baseline to Week 12
  Change in self-reported cigarettes smoked daily

SECONDARY OUTCOMES:
Subjective response to an e-cigarette | From Baseline to Week 12
  To assess subjective satisfaction and other perceived rewarding or aversive effects accompanying e-cigarette use and combustible cigarette use using the modified (e-Cigarette) Cigarette Evaluation Questionnaire. This questionnaire contains five subscale scores: smoking satisfaction (satisfying, tastes good, enjoy smoking), psychological rewards (calms down, more awake, less irritable, helps concentrate, reduces hunger), aversion (dizziness, nauseated), enjoyment of respiratory tract sensations (single-item assessment), craving reduction (single-item assessment). Participants will be asked to assess the 12 items of the questionnaire on a 7-point scale, ranging from "not at all" to "extremely".

OTHER OUTCOMES:
Number of participants that completely switch from combustible cigarettes to e-cigarette | Daily during Week 9 - Week 12
  Self-report of no smoking
Number of participants that completely switch from combustible cigarettes to e-cigarette | Week 9 - Week 12
  Expired air carbon monoxide (CO) value of <5 ppm
Number of participants that completely switch from combustible cigarettes to e-cigarette | Week 12
  Expired air carbon monoxide (CO) value of <5 ppm
Number of participants that completely switch from combustible cigarettes to e-cigarette | Week 12
  Self-report of no smoking

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rose Research Center, Charlotte, North Carolina
  - Rose Research Center, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rose JE, Behm FM, Cohen G, Willette PN, Botts TL, Botts DR. Smoking reduction using an electronic nicotine delivery system (ENDS) with nicotine delivery similar to combustible cigarettes. Harm Reduct J. 2024 Jul 29;21(1):142. doi: 10.1186/s12954-024-01064-0. PMID 39075535